CLINICAL TRIAL: NCT01435850
Title: "Enfoncement de la Tige SL-PLUS et de la Tige SL-PLUS MIA:Etude Comparative"
Brief Title: Safety and Efficacy of the SL PLUS and the SL PLUS MIA Hip Stem
Acronym: SL-PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: D10056-2-F
Record Dates: First submitted 2011-09-13; First posted 2011-09-19 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Coxarthrosis
Keywords: hip arthroplasty; primary stability; secondary stability; EBRA
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIP STEM SL PLUS (Sham Comparator): study group
  Interventions: Procedure: primary total hip arthroplasty
- HIP STEM SL PLUS MIA (Active Comparator): control group
  Interventions: Procedure: primary total hip arthroplasty

INTERVENTIONS:
Procedure: primary total hip arthroplasty — All patients eligible to the study criteria will be included. A total hip arthroplasty unilateral will be performed.
  Other Names: SL-PLUS, SL-PLUS MIA, Lateralized hip stem

SUMMARY:
Randomized controlled trial using two types of hip stems, SL PLUS MIA (control group) and SL PLUS (study group).

We compare primary and secondary stability of both hip stems for radiographic outcome using EBRA (Ein-Bild-Roentgen-Analyse) after a two year follow-up period.

Further, we compare all differences in clinical outcome using Harris Hip Score, Oxford hip score and radiographic findings.

DETAILED DESCRIPTION:
This study is a monocentric study, randomized and controlled including two types of hip stems: SL PLUS MIA (control group) and SL PLUS (study group).

Each group will include 45 patients where a number of 5 patients for each group calculated extra in case of loss.

Patients will be followed after

* 6 weeks
* 6 months
* 12 months
* 24 months. Radiographs are taken in a-p and lateral view using a standard protocol. Primary and secondary stability of both hip stems will be analyzed using the EBRA software (Ein-Bild-Roentgen-Analyse, University of Innsbruck, Austria) after the completion of the two year follow-up.

Further, we compare all differences in clinical outcome using Harris Hip Score, Oxford hip score and radiographic findings such as radiolucent lines.

ELIGIBILITY:
Inclusion Criteria:

* Patient needs primary total hip arthroplasty with SL-PLUS (standard or lateralized depending on bone morphology)
* Age at surgery : 18-80 years old
* Patient has social security number
* Patient gives Informed Consent (IC) by signing the IC form and patient is willing to attend the follow-up control

Exclusion Criteria:

* Patient's BMI is over 35
* Patient has bone tumors that can affect implant stability
* Patient needs cortical steroid treatment
* Patient needs hip revision arthroplasty
* Patient has general inflammation that could affect bone quality
* Patients classified Charnley C

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2012-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Stability of primary total hip arthroplasty | 24 months
  Study compares the stability of two types of hip stems using the Femoral Component Analysis (FCA-EBRA)method. 4 images of a-p pelvic view will be collected over a 2-year period: at 6 weeks, 6, 12 and 24 months.

SECONDARY OUTCOMES:
Oxford Hip Score | 24 months
  According to Delaunay C, Cross-cultural adaptations of the Oxford-12 HIP score to the French speaking population, Orthop Traumatol Surg Res. 2009 Apr;95(2):89-99. Epub 2009 Apr 3.
  Oxford Hip Score will be measured pre-operatively, after 6 weeks, 6, 12 and 24 months.
Harris Hip Score | 24 months
  Harris Hip Score will be measured pre-operatively, after 6, 12 and 24 months. No measurement after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Henri Migaud, MD, Pr., Principal Investigator — University Hospital
Locations (1):
- Hopital Salengro, Service d'Orthopédie C, Lille, France